CLINICAL TRIAL: NCT00283660
Title: Zinc, Mental Health, and School Performance
Brief Title: Zinc, Mental Health, and School Performance in Guatemalan Schoolchildren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Institute of Nutrition of Central America and Panama (INCAP) (Unknown); Mexican National Institute of Public Health (Other Government)
Responsible Party: Principal Investigator, Aryeh David Stein, Professor, Global Health, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00045755; R01MH067981 (NIH); DSIR 84-CTM
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Depression; Anxiety
Keywords: Zinc; Dietary Supplements; Nutritional Supplements; Child; Mental Health; School; Guatemala
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being | interventions — Zinc Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): Dietary Supplement: 10 mg zinc oxide
  Interventions: Dietary Supplement: 10 mg zinc oxide
- Placebo (Placebo Comparator): Placebo (double blinded)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: 10 mg zinc oxide — 10 mg zinc oxide
  Arms: Active
Other: Placebo — Placebo pill taken five days a week for six months.
  Arms: Placebo

SUMMARY:
This study will determine whether supplements of the mineral zinc will improve mental health and school performance among schoolchildren in Guatemala.

DETAILED DESCRIPTION:
Mental health problems are an important cause of dysfunction throughout the world, accounting for 8.1% of the Global Burden of Disease. The need for interventions that can prevent mental health conditions, particularly among children, cannot be overemphasized. This study will determine whether zinc supplementation improves the mental health and school performance among children in Guatemala.

Participants will be randomly assigned to receive daily supplements of either zinc or placebo for 6 months. Participants will be assessed at study entry and after the 6-month treatment. Participants and their parents and teachers will complete questionnaires about the participants' symptoms of depression and anxiety, concentration and activity levels, school performance, and any environmental stressors to which the participants may be exposed to.

ELIGIBILITY:
Inclusion Criteria:

* Attend a public school in specific Guatemalan community and has thorough and up-to-date school records
* Currently in 2nd to 6th grade
* Parent or guardian willing to provide informed consent

Exclusion Criteria:

* Any illness that may affect participants' zinc levels
* Any chronic illness
* History of cancer

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 750 (Actual)
Dates: Start 2006-01; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Symptoms of depression | Baseline and post supplementation

SECONDARY OUTCOMES:
Symptoms of anxiety | Baseline and post supplementation
attention problems and school performance | Baseline and post supplementation
activity levels | Baseline and post supplementation
zinc levels | Baseline and post supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Aryeh D Stein, PhD, Principal Investigator — Emory University
Locations (1):
- Instituto de Nutrición de Centro América y Panamá - INCAP, Guatemala City, Guatemala

REFERENCES:
- [Result] DiGirolamo AM, Ramirez-Zea M, Wang M, Flores-Ayala R, Martorell R, Neufeld LM, Ramakrishnan U, Sellen D, Black MM, Stein AD. Randomized trial of the effect of zinc supplementation on the mental health of school-age children in Guatemala. Am J Clin Nutr. 2010 Nov;92(5):1241-50. doi: 10.3945/ajcn.2010.29686. Epub 2010 Sep 29. PMID 20881069
- [Result] Bui VQ, Stein AD, DiGirolamo AM, Ramakrishnan U, Flores-Ayala RC, Ramirez-Zea M, Grant FK, Villalpando S, Martorell R. Associations between serum C-reactive protein and serum zinc, ferritin, and copper in Guatemalan school children. Biol Trace Elem Res. 2012 Aug;148(2):154-60. doi: 10.1007/s12011-012-9358-0. Epub 2012 Feb 22. PMID 22354676